CLINICAL TRIAL: NCT04322695
Title: A Rehabilitation Education Care Program on Return to Work Among Head and Neck Cancer Survivors - Improve Disability and Barriers of Return to Work
Brief Title: A Rehabilitation Education Care Program on Return to Work Among Head and Neck Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Shu-Ching Chen, Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201801245B0
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Education Care Program (RECP) (Experimental): Cancer rehabilitation program and patients education can improve disability and promote return to work.
  Interventions: Behavioral: Rehabilitation Education Care Program
- Usual care (Other): Usual care
  Interventions: Behavioral: Rehabilitation Education Care Program

INTERVENTIONS:
Behavioral: Rehabilitation Education Care Program — The RECP contained the following domains: (1) assessment and detection of disability; (2) home exercise; (3) activities to improve mobility; (4) dietary management; (5) patient education; and (6) vocational counseling.

SUMMARY:
The purpose of this study will to identify factors (performance ability, physical function, psychosocial function, fear of cancer progression, social support, demographic characteristics, and disease-related characteristics) that impact the Return to work and work status in survivors of HNC within one year after completion treatment. Head and neck cancer survivors who have attended a rehabilitation education care program (RECP) intervention will have better performance ability, physical function, psychosocial function, fear of cancer progress, social support, and lower return to work to patients who not attended with the intervention.

DETAILED DESCRIPTION:
The purpose of this 2-year project will involve a randomized controlled clinical trial to evaluate the 3-months RECP. Eligible participants will be recruited from initial completion treatment to 6 months after completion treatment and randomized into a control group and an experimental group, with the control group patients receiving routine hospital care and the experimental group patients receiving the 3-months RECP. Outcomes will be assessed using Return to Work Barrier Scale (RTWBS), Fear of Progression Questionnaire (FoP-Q-SF), Social Support Scale (SSS), University of Washington Quality of Life Scale (UW-QOL), Karnofsky's Performance Score (KPS), Katz Activities of Daily Living Scale (ADL), and Instrument Activities of Daily Living Scale (IADL). Subjective data will be collected at four time points: baseline (6 months after completion of treatment)(T0) and then 9, 12, and 18months after completion of treatment (T1, T2, and T3, respectively). Objective data will be assessed at the same time points. The mixed-model repeated measure ANOVA will be used to analyze the data. The investigators plan to recruit 30 subjects for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of head and neck cancer.
2. Must be age were greater than 18 years and less than 64.5 years
3. Must be able to better performance status and KPS score more than 60
4. Must be had completion of treatment more than 3 months

Exclusion Criteria:

1. Unemployment or retire at the time of cancer diagnosis
2. unstable systemic disease
3. Poor performance status and KPS score less than 60

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change barrier to return to work | 3 months, 6 months, and 12 months
  Return to Work Barrier Scale (RTWBS)

SECONDARY OUTCOMES:
Change fear of cancer progress | 3 months, 6 months, and 12 months
  Fear of Progression Questionnaire (FoP-Q-SF)
Change social support | 3 months, 6 months, and 12 months
  Social support/Social Support Scale (SSS)
Change quality of life | 3 months, 6 months, and 12 months
  University of Washington Quality of Life Scale (UW-QOL)

CONTACTS AND LOCATIONS:
Locations (1):
- Shu-Ching Chen, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chang YL, Huang BS, Lin CY, Chung CF, Chen SC. Effects of a return to work program on the health and barriers to returning to work in head and neck cancer patients: A randomized controlled trial. Asia Pac J Oncol Nurs. 2023 Oct 17;10(12):100320. doi: 10.1016/j.apjon.2023.100320. eCollection 2023 Dec. PMID 38059206